CLINICAL TRIAL: NCT06749925
Title: Phase III Randomized, Double-Blind, Placebo-Controlled Clinical Trial Assessing the Efficacy and Safety of Dendritic Cell-Based Immunotherapy for Glioblastoma
Brief Title: Clinical Trial Assessing the Efficacy and Safety of Dendritic Cell-Based Immunotherapy for Glioblastoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Jose Alexandre Marzagão Barbuto, Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 58882116.7.3001.0065
Record Dates: First submitted 2024-11-22; First posted 2024-12-27 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Glioblastoma
Keywords: glioblastoma; dendritic cell; vaccine; clinical trial
MeSH Terms: conditions — Glioblastoma | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- DC Vaccine Arm (Experimental): This group is receiving the dendritic cell vaccine.
  Interventions: Biological: Dendritic Cell Vaccine
- DC Vaccine + Pembrolizumab Arm (Active Comparator): This group is receiving the dendritic cell vaccine combined with pembrolizumab.
  Interventions: Combination Product: Pembrolizumab
- Placebo Control Arm (Placebo Comparator): This group is receiving a placebo and serves as the control.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Dendritic Cell Vaccine — This intervention distinguishes itself from others by utilizing allogeneic dendritic cells derived from healthy donors fused with autologous tumor cells from patients, which is a novel approach compared to the commonly used autologous DC-based vaccines (DCVax).
  Arms: DC Vaccine Arm
Combination Product: Pembrolizumab — Recent findings have shown that the anti-PD1 monoclonal antibody, a checkpoint inhibitor, can sustainably enhance the anti-tumor immune response. In this study, all patients in the intervention group (vaccine) who reach the fifth dose will be randomized to receive either pembrolizumab or a placebo as an addition to the experimental treatment regimen.
  Arms: DC Vaccine + Pembrolizumab Arm
Other: Placebo — In this study, all patients in the intervention group (vaccine) who reach the fifth dose will be randomized to receive either pembrolizumab or a placebo as an addition to the experimental treatment regimen.
  Arms: Placebo Control Arm

SUMMARY:
This Phase III, multicenter, placebo-controlled clinical trial with sequential randomization is designed to evaluate the efficacy and safety of an experimental vaccine composed of hybrid dendritic cells (DCs) for the treatment of glioblastoma. Conducted at the Hospital das Clínicas of the University of São Paulo Medical School (HCFMUSP) and the Institute of Biomedical Sciences of the University of São Paulo (ICB/USP), the study is led by Professor José Alexandre Marzagão Barbuto. A multidisciplinary team of researchers specializing in neurosurgery, pathology, hematology, and other fields will contribute to a comprehensive approach.

The trial aims to determine whether the hybrid DC vaccine can increase overall survival in adult patients with glioblastoma who have completed standard treatment, including surgery, chemotherapy, and radiotherapy. Secondary objectives include evaluating progression-free survival, quality of life, immune response, and the safety of the intervention. The study will enroll 186 patients, who will be randomized into three groups: (1) a control group receiving placebo, (2) a group receiving the DC vaccine, and (3) a group receiving the DC vaccine combined with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a histological diagnosis of glioblastoma and confirmed IDH status.
* Currently undergoing standard-of-care treatment, which includes surgery, chemotherapy, and radiotherapy.
* Availability of pre-treatment magnetic resonance imaging (MRI).
* Ability to attend clinical follow-ups every 2 months.
* Functional performance score > 50 at the time of study enrollment.
* Tumor cells capable of expansion in culture.

Exclusion Criteria:

* Patients with any concomitant neoplasm (except basal cell carcinoma).
* Pregnant or breastfeeding individuals.
* Patients with significant medical or surgical conditions as determined by the study team, psychiatric disorders, or those requiring medications or treatments that could interfere with study procedures or the evaluation of the vaccine's safety and efficacy.
* Patients who are HIV-positive, immunosuppressed, and/or have undergone organ transplantation.
* Refusal or inability to provide consent, such as patients with aphasia.
* Participation in any experimental treatment protocols within the 6 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From enrollment to the end of treatment at 2 years
  The primary expected outcome is overall survival, evaluated over a 2-year period.

SECONDARY OUTCOMES:
Disease Progression and Survival Metrics | From enrollment to the end of treatment, limited to 2 years
  Progression-free survival in months, assessed through RANO criteria (complete response, partial response, stable disease or progressing disease); Survival rates at 6 and 12 months after the initiation of vaccination; Functional status evolution, evaluated through the Karnofsky Performance Scale (KPS, ranging from 0, dead to 100, asymptomatic), WHO-ECOG scale (Eastern Cooperative Oncology Group, ranging from 0, fully active, to 5, dead), and Mini-Mental State Examination (MMSE, ranging from 0, all questions responded wrongly to 30, best performance);
Quality of life and general health assessment | From enrollment to the end of treatment, limited to 2 years
  Quality of life and general health evaluation:
  FACT-Br (Functional Assessment of Cancer Therapy - Brain / 5 point Likert-type scale ranging from 0 "not at all" to 5 "very much") BCM-20 (Brain Cancer Module-20) MDASI-BT (MD Anderson Symptom Inventory for brain tumor / assesses the severity of symptoms at their worst in the last 24 hours on a 0-10 NRS, with 0 being "not present" and 10 being "as bad as you can imagine.") EORTC-QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 / Likert scale ranging from 0 "not at all" to 4 or 7 "very much") EORTC QLQ-BN20 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Brain Neoplasm 20 / 4 point Likert-type scale ranging from 0 "not at all" to 4 "very much") EQ-5D-5L (European Quality of Life 5 Dimensions 5 Level Version / scale ranging from level 1: no problems to Level 5: extreme problems)
Immunological Response | From enrollment to the end of treatment, limited to 2 years
  Levels of Th1-pattern tumor-reactive T lymphocytes in peripheral blood.
Safety Profile | From enrollment to the end of treatment, limited to 2 years
  Adverse events classified according to the U.S. National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (2010).

IPD SHARING:
Plan to Share IPD: Undecided